CLINICAL TRIAL: NCT04055233
Title: Reduction of Postoperative Wound Infections by Antiseptica?
Acronym: RECIPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johannes Lauscher (Other)
Responsible Party: Sponsor-Investigator, Johannes Lauscher, Principal investigator, MD, PhD, Staff surgeon, Department of General, Visceral and Vascular Surgery, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-001551-22
Record Dates: First submitted 2018-04-25; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — polihexanide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two arm prospective randomized single center interventional trial. 1:1 randomization into experimental arm (irrigation with polyhexanide) and control arm (irrigation with saline).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous irrigation with 0.04% polyhexanide solution (Experimental): Intervention: after closure of abdominal fascia, an intraoperative irrigation of the subcutaneous tissue with 250 ml antiseptic solution (0.04% polyhexanide) will be done once for ten minutes.
  No subcutaneous suture. Closure of skin with either staples, interrupted sutures or running suture.
  Interventions: Drug: Polihexanide; Serasept
- Subcutaneous irrigation with NaCl (saline) (Active Comparator): Intervention: after closure of fascia, an intraoperative irrigation of the subcutaneous tissue with 250 ml NaCl (saline) will be done once for one minute.
  No subcutaneous suture. Closure of skin with either staples, interrupted sutures or running suture.
  Interventions: Drug: NaCl; saline

INTERVENTIONS:
Drug: Polihexanide; Serasept — Experimental arm: irrigation of subcutaneous tissue after fascia closure with polihexanide (ten minutes).
  A single dose of perioperative antibiotics (cefuroxim alone or cefuroxim and metrodidazole in bowel surgeries) was given 30 minutes before skin incision.
  Hair removal was done with electronic clippers and preoperative skin antisepsis was performed with propanol and povidone-iodine.
  Before closure of fascia, instruments and gloves were changed. No subcutaneous suture was used. Skin was closed either with skin staples, continuous intracutaneous suture or interrupted suture.
  All surgeries were done according to the Standard Operating Procedures of the Department for General, Visceral and Vascular Surgery, Charité Campus Benjamin Franklin.
  Other Names: Polihexanide (0.04% antiseptic solution)
  Arms: Subcutaneous irrigation with 0.04% polyhexanide solution
Drug: NaCl; saline — Control arm: irrigation of subcutaneous tissue after fascia closure with NaCl (one minute) A single dose of perioperative antibiotics (cefuroxim alone or cefuroxim and metrodidazole in bowel surgeries) was given 30 minutes before skin incision.
  Hair removal was done with electronic clippers and preoperative skin antisepsis was performed with propanol and povidone-iodine.
  All surgeries were done according to the Standard Operating Procedures of the Department for General, Visceral and Vascular Surgery, Charité Campus Benjamin Franklin.
  Before closure of fascia, instruments and gloves were changed. No subcutaneous suture was used. Skin was closed either with skin staples, continuous intracutaneous suture or interrupted suture.
  All surgeries were done according to the Standard Operating Procedures of the Department for General, Visceral and Vascular Surgery, Charité Campus Benjamin Franklin.
  Other Names: NaCl (saline)
  Arms: Subcutaneous irrigation with NaCl (saline)

SUMMARY:
Wound infections are a frequent complication in abdominal surgery. The investigators hypothesize that the antiseptic solution 0.04 % polyhexanide (serasept) may reduce occurrence of postoperative wound infections compared to NaCL (saline) solution in a prospective randomized setting.

DETAILED DESCRIPTION:
Invstigator initiated monocenter randomized controlled trial. Intraoperative irrigation of subcutaneous tissue with NaCl (saline) solution or antiseptic solution 0.04 % polyhexanide (Serasept) in elective abdominal surgery. Primary endpoint: SSI 30 days postoperatively according to CDC criteria.

ELIGIBILITY:
Inclusion Criteria: - planned laparotomy for visceral surgery

Exclusion Criteria:

* Age under 18 years
* allergy against polihexanid
* laparoscopic surgery
* emergency surgery
* lack of understanding of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
surgical site infection | 30 days postoperatively
  Surgical site infection according to CDC definition.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes C Lauscher, MD, Principal Investigator — Charité-University Medicine (Berlin, Germany)
Locations (1):
- Charité Campus Benjamin Franklin, Steglitz, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strobel RM, Leistner R, Leonhardt M, Neumann K, Eschlbock SM, Lee LDG, Seifarth C, Schineis CHW, Kamphues C, Weixler B, Beyer K, Lauscher JC. Is There an Association between Intra-Operative Detection of Pathogens in Subcutaneous Tissue and Surgical Site Infections? Results from a Prospective Study. Surg Infect (Larchmt). 2022 May;23(4):372-379. doi: 10.1089/sur.2021.154. Epub 2022 Mar 9. PMID 35263172
- [Derived] Strobel RM, Leonhardt M, Krochmann A, Neumann K, Speichinger F, Hartmann L, Lee LD, Beyer K, Daum S, Kreis ME, Lauscher JC. Reduction of Postoperative Wound Infections by Antiseptica (RECIPE)?: A Randomized Controlled Trial. Ann Surg. 2020 Jul;272(1):55-64. doi: 10.1097/SLA.0000000000003645. PMID 31599810